CLINICAL TRIAL: NCT06175858
Title: Validation of Different Diagnostic Modalities in the Detection of Cardiac Amyloidosis Among Patients With "Red Flags"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alsayed Ali Mahmoud Ahmed, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cardiac amyloidosis
Record Dates: First submitted 2023-11-22; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population with echocardiographic or clinical red flags for cardiac amyloidosis (Other): The study aims at including all population with the previously described red flags
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: CMR — We will use cmr and bone scintigraphy to detect cardiac amyloidosis due t the high accuracy and reliability
  Other Names: BONE SCINTIGRAPHY

SUMMARY:
The study aims to test and compare the diagnostic yield of different diagnostic modalities (speckle tracking echocardiography, CMR, serum and urine protein analysis and bone tracer scintigraphy) in the detection of cardiac amyloidosis among patients with "red flags" suspecting cardiac amyloidosis.

DETAILED DESCRIPTION:
Cardiac amyloidosis (CA) is a condition that can be caused by rare genetic variants in the hereditary forms or because of acquired conditions. It is one of the serious and progressive infiltrative disease that is caused by the deposition of amyloid fibrils at the cardiac level .

Cardiac amyloidosis causes restrictive cardiomyopathy, and this is caused by extracellular deposition of proteins in the myocardium. The proteins have an unstable structure that causes them to misfold, aggregate, and deposit as amyloid fibrils .

According to the nature of the infiltrating protein, cardiac amyloidosis has two main subtypes, immunoglobulin light chain cardiac amyloidosis (AL-CA), and transthyretin cardiac amyloidosis (ATTR-CA) which is further subdivided according to the presence or absence of a mutation in the transthyretin gene into wild-type (ATTRwt-CA) and variant (ATTRv-CA) .

Despite of being one of the most serious, fetal diseases, and a considerable cause of heart failure with preserved ejection fraction (HFpEF), cardiac amyloidosis is still significantly underdiagnosed, this may be due to its varied presentations and lack of awareness about the nature of the disease. Awareness of "red flags" suggestive of amyloidosis can enhance one's index of appropriate clinical suspicion and enable earlier diagnosis of CA .

Diagnosis of CA:

Diagnosis and classification of CA needs high index of clinical suspicion and awareness of clinical clues suggestive of CA. This ranges from ECG, echocardiography, speckle tracking, laboratory investigations, bone scan scintigraphy and cardiac MRI.

ECG:

Although ECG may be normal even at advanced stages of CA, it can provide clues for amyloid infiltration and further support the diagnosis in conjunction with imaging findings. The typical finding is normal or low QRS voltage (<1 mV in the precordial and <0.5 mV in the extremity leads) in patients with LV hypertrophy on echocardiography. This is more common in AL-CA (45%) but less frequent in ATTR-CA (23-31%) .

Other features include pseudo-infarct pattern with Q waves or slow R-wave progression in the precordial leads, atrioventricular block or bundle branch block. Atrial fibrillation is the most common arrhythmia with a high relapse rate .

Echocardiography:

1. Conventional Measures and Diastolic Function Transthoracic echocardiography is usually the initial imaging technique for evaluating patients with suspected cardiac amyloidosis. Typical echocardiographic findings are increased left ventricular (LV) wall thickness over 12 mm, accompanied by additional thickening of the right ventricle (RV), valves, and interatrial septum, and generally small pericardial effusion .

   Furthermore, bi-atrial dilatation is frequently observed in severe diastolic dysfunction. The characteristic speckled appearance of the myocardium, on the other hand, referred to as "granular sparkling," has been described in patients with cardiac amyloidosis and previously deemed as a key factor in establishing the diagnosis .

   However, granular sparkling can also be present in other causes of LV hypertrophy, yielding lower sensitivity for identifying cardiac amyloidosis than previously anticipated. In addition, tissue harmonic imaging and image processing techniques may alter the myocardial echogenicity and, thus, impair the diagnostic value of this feature .

   Generally, LV diastolic abnormalities occur already in the early stages of cardiac amyloidosis. In contrast, LV ejection fraction usually remains normal or mildly reduced until the late stages of the disease, despite diminished longitudinal deformation of the myocardium. Despite preserved ejection fraction, cardiac output is low due to decreased ventricular volumes .

   In this regard, myocardial contraction fraction, the ratio of (LV) stroke volume to myocardial volume measured by M-mode echocardiography, was predictive of mortality in patients with ATTRv, ATTRwt, and AL amyloidosis .
2. The Role of Echocardiographic Myocardial Deformation (Strain) Changes in the myocardium in dimensions and shape during contraction and relaxation can be characterized by assessing myocardial "strain." Strain is a measure of regional or global deformation, which originates from physics and can be applied to the heart to measure regional shortening, thickening, and lengthening of the myocardium. Strain can be quantitatively assessed by echocardiography using speckle tracking imaging and has demonstrated a characteristic pattern with markedly reduced strain in mid and basal and relatively preserved strain in apical segments. This pattern is referred to as "apical sparing" and is well suited for differentiating such patients from other causes of LV hypertrophy (13). The apical sparing pattern is easily recognizable on polar myocardial strain maps and is observed in patients with ATTR and AL cardiac amyloidosis.

In addition, in several previous clinical studies, the myocardial strain was shown to bear prognostic implications in amyloidosis, exhibiting incremental value over clinical and biochemical markers for the risk stratification of patients with AL amyloidosis .

Laboratory testing:

As no single parameter exists for diagnosing ATTR-CA, the goal of laboratory testing in patients with suspected CA is primarily to search for markers of plasma cell disease causing AL-amyloidosis. These include elevated serum free light chain immunoglobulins, pathologic to free light chain ratio and monoclonal gammopathy in serum and urine immunofixation with reported sensitivity of >95% for the detection of AL amyloidosis .

Urine protein analysis can also be helpful in diagnosis cardiac amyloidosis and differentiating the type.

Bone Tracer Scintigraphy:

Cardiac uptake of 99mTc-phosphate derivatives was first demonstrated in the 1980s as an accidental finding in patients with ATTR- CA undergoing scintigraphy for metastatic bone disease. In 2005 a small study demonstrated the diagnostic value of 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD) for ATTR-CA .

Since then, several studies reported on the high sensitivity of bone-tracer scintigraphy for ATTR-CA with only mild or absent tracer uptake in AL-CA, attributed possibly to higher calcium con- tent in ATTR amyloid deposits .

These results were recently validated in a large-scale multicenter trial, which showed high diagnostic accuracy of 99mTc-phosphate scintigraphy for non-invasive detection of ATTR-CA .

Qualitative visual Perugini scale relate heart uptake as compared with rib bone uptake and include grade 0 = no uptake, grade 1 = mild uptake, less than rib (less than bone for 99mTc-DPD), grade 2 = moderate uptake, equal to rib, grade 3 = severe uptake, greater than rib.

In summary, a scan demonstrating grade 2 or 3 uptake according to the visual Perugini scale combined with negative serum and urine analysis for elevated free light chains and monoclonal gammopathy demonstrated 99% sensitivity, 100% positive predictive value and 100% specificity for ATTR-CA .

Cardiac Magnetic Resonance (CMR):

1. Conventional Cine Measures by CMR:

   CMR allows for non-invasive imaging of cardiac structures with high spatial resolution and intrinsic blood-to-tissue contrast. The versatility of CMR can provide the assessment of myocardial function, perfusion, tissue characterization by late gadolinium enhancement (LGE) and mapping techniques, and, if required, myocardial deformation using "strain" analyses within a single examination, independent of the patients' acoustic windows and without radiation exposure .

   Morphological and functional alterations are comparable with echocardiography findings. In addition, CMR studies highlighted differences in asymmetrical septal hypertrophy in ATTR amyloidosis, mimicking hypertrophic cardiomyopathy versus concentric hypertrophy seen in most patients with AL amyloidosis .
2. Late Gadolinium Enhancement:

   Gadolinium is an extracellular contrast agent. Therefore, gadolinium distributes preferentially in areas of increased extracellular volume (ECV), as in diseased myocardium with an expanded extracellular space in patients with cardiac amyloidosis. In contrast, the contrast agent rapidly washes out in healthy myocardium. LGE images are typically acquired approximately 10 min after contrast agent administration. LGE allows for visual and if required, quantitative assessment of the myocardial amyloid burden, albeit challenging in diffuse global LGE with progressed disease cases. Several studies previously demonstrated the presence of LGE in patients with cardiac amyloidosis .

   The sensitivity and specificity of LGE versus endomyocardial biopsy for diagnosing cardiac amyloidosis were reported to be 86% and 92%, respectively, based on a recent meta-analysis .
3. Native T1 Mapping and Extracellular Volume (ECV):

Native T1 Measures of the myocardial T1 relaxation with non-contrast T1 mapping sequences have been used to detect and quantify interstitial expansion due to fibrosis . In cardiac amyloidosis, native T1 mapping exhibited significantly higher values in patients than in control subjects. In the same direction, T1 elevations were noted in AL and ATTR amyloidosis patients, allowing for differentiation between both subtypes of amyloidosis versus hypertrophic cardiomyopathy with high accuracy . In addition, native T1 values were shown to be related to functional echocardiographic markers of systolic and diastolic LV function and significantly increased even in asymptomatic amyloidosis patients, thus being potentially more sensitive than LGE .

Extracellular Volume (ECV) By measuring the T1 value of the myocardium before and after gadolinium administration, the myocardial ECV can be quantified. This parameter reflects the fraction of myocardium composed by the extracellular space, where the amyloid deposits accumulate in patients with cardiac amyloidosis. ECV requires administering gadolinium-based contrast agents but is less susceptible to technical issues than the pulse sequences used for native T1 mapping . Like native T1, ECV has been extensively validated in cardiac amyloidosis , including studies where ECV was serially studied during treatment with novel pharmacologic agents in AL and ATTR amyloidosis. Due to its high reproducibility and quantitative nature, the use of ECV was proposed for serial studies, monitoring the response to therapies in patients with cardiac amyloidosis. In addition, ECV has been validated against histology, exhibiting a close correlation to histologic amyloid burden and was independently associated with patients' outcomes .

In ATTR amyloidosis, ECV was, in contrast to native T1 values, independently associated with mortality after adjustment for age, biochemical, functional markers, and LGE. This highlights the robustness of this marker which was recently confirmed in a meta-analysis by a systematic comparison of ECV versus native T1 in AL and ATTR amyloidosis patient cohorts. Summarizing the relevance of native T1 and ECV, both markers bear diagnostic solid and prognostic implications and need to be considered together with clinical, laboratory, and other imaging parameters during the diagnostic work-up of patients with suspected cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* "Red flags" include any one of the following:

Clinical "Red flags":

* Bilateral carpal tunnel syndrome (30).
* "Popeye sign", rupture of long head of the biceps tendon.
* Lumbar spinal canal stenosis in association with unilateral carpal tunnel syndrome (31).

Echocardiographic/imaging "Red Flags"

* LV wall thickness ≥ 12 mm and heart failure in men > 60 y/ women > 70y.
* LV wall thickness ≥ 12 mm and AV-Block or pacemaker.
* Infiltrative phenotype (biventricular hypertrophy, thickening of cardiac valves, pericardial effusion, thickening of the interatrial septum).
* LV wall thickness ≥ 12 mm and low voltage on ECG.
* Paradoxical low flow/low gradient aortic stenosis.

Exclusion Criteria:

- 1. Patient who refuse to give a consent to the following investigations. 2. Patient with any contra-indication to undergo CMR, or bone scintigraphy will be excluded e.g., non compatible implantable cardiac devices, claustrophobic, severe kidney function impairment.

3. Patient with established diagnosis of other infiltrative cardiac disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Validation of different diagnostic modalities in the detection of cardiac amyloidosis among patients with "red flags" | Baseline
  • Detect the diagnostic yield of different diagnostic modalities for detection of cardiac amyloidosis and compare them.

SECONDARY OUTCOMES:
i. Identification of the percentage of patients who will have a final confirmed diagnosis of cardiac amyloidosis among all included patients with "red flags". | Baseline
  j. Identification of the most sensitive and specific "red flag" or combination of "red flags" to detect cardiac amyloidosis.